CLINICAL TRIAL: NCT05984563
Title: Official Title Optimization Strategy to Predict and Individualize Oxygen Delivery During Cardiac Surgery Under Cardiopulmonary Bypass
Brief Title: Optimization Strategy for Oxygen Delivery Under Cardiopulmonary Bypass
Acronym: OPTI-DO2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0705
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Surgery
Keywords: Oxygen delivery; Cardiopulmonary bypass; Cardiac surgery; Goal-directed perfusion; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cardiopulmonary bypass — CPB will be ensured as usual care: priming volume will be set as 1200 to 1500 mL. Patient blood management and hemodynamic management will be left at the discretion of the anesthesiologist in charge of the patient. Anticoagulation during CPB will be handled through an initial heparin bolus of 300-400 UI/kg followed by additional boluses to maintain ACT above 400 s. Non-heparin-coated bypass circuits incorporating an integrated phosphorylcholine-coated oxygenation system will be used.

SUMMARY:
Cardiac surgery is a frequent procedure that can lead to serious complications, including acute kidney injury (AKI) or postoperative delirium. During the intervention, a cardiopulmonary bypass (CPB) is used to ensure tissue perfusion and oxygen delivery (DO2). The hypothesisis that an individualized strategy to optimize DO2 during CPB could decrease complications rate after cardiac surgery. Indeed, it is known that DO2 depends on CPB output, hemoglobin level and O2 tension. To this day, a DO2 threshold below 280 mL is known to be associated with postoperative AKI. From these data, a "Goal Directed Perfusion" strategy is widely used to maintain a DO2 above this threshold during CPB. But DO2 decrease in unpredictable, and the other factors influencing DO2 interindividual variability are not known. Moreover, the relation between DO2 and tissue perfusion is not well established, as DO2 requirement could differ between individuals or organs. Population approach using nonlinear mixed models is a method used to optimize drug administration with pharmacokinetics and pharmacodynamics models. Using this method, the aim of this study is to evaluate DO2 variability during CPB and develop a model to optimize GDP strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* Patients scheduled for elective cardiac surgery under CPB at the university hospital of Lille, France
* Patients with given written consent
* Patient insured under the French social security system

Exclusion Criteria:

* Pregnant or breastfeeding
* Off pump cardiac surgery
* Lack of DO2 monitoring
* Emergency surgery (infectious endocarditis, aortic dissection, cardiac transplantation, LVAD implantation) Uncontrolled sepsis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery under CPB at the university hospital of Lille, France
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-24 (Estimated); Study Completion 2024-04-04 (Estimated)

PRIMARY OUTCOMES:
values oF D02 calculated with the CONNECT software (LivaNova, London, United Kingdom) using CPB output and hemoglobin values (measured using Spectrum Medical M4) (standard care) | Every 20 to 30 seconds during CPB (standard care) and up to 28 days

SECONDARY OUTCOMES:
Incidence of postoperative AKI using creatinine measurement (standard care) | up to 48 hours postoperative
Incidence of postoperative deliriumassessed by CAM-ICU, CPC and mRS scores | up to 48 hours postoperative
Vital status checklist | up to 28 days postoperative